CLINICAL TRIAL: NCT04914507
Title: A Prospective Analysis of Long-Term Clinical Outcomes and 3D Spine Growth in Anterior Vertebral Body Tethering
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Pediatric Spine Foundation (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PSSG0121
Record Dates: First submitted 2021-05-31; First posted 2021-06-04 (Actual); Last update posted 2023-11-15 (Actual); Status verified 2023-11

CONDITIONS: Scoliosis Idiopathic
Keywords: anterior vertebral body tethering

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Anterior Vertebral Body Tethering (Other): The subject is will receive anterior vertebral body tethering surgery, as clinically indicated, after all pre-operative assessments are complete.
  Interventions: Device: Anterior Vertebral Body Tethering

INTERVENTIONS:
Device: Anterior Vertebral Body Tethering — Subject will receive anterior vertebral body tethering surgery.

SUMMARY:
Anterior vertebral body tethering (AVBT) is a novel, minimally invasive, growth modulation technique that was recently approved by the FDA under a Humanitarian Device Exemption (HDE). The goal of AVBT is to control curve progression by applying compression on the convex side of the spine deformity. While there has been great initial enthusiasm about the technique as an alternate treatment option to spinal fusion for skeletally immature children with scoliosis, there is a need to better understand the long-term outcomes.

The purpose of this study is to report the long-term clinical outcomes of skeletally immature patients treated with AVBT, specifically:

1. The effect on three-dimensional spine growth as compared to normal controls
2. Maintenance of major Cobb angle less than or equal to 50 degrees at skeletal maturity
3. Complications associated with both the procedure and the device

ELIGIBILITY:
Inclusion Criteria: Skeletally immature patients that receive AVBT surgical treatment to obtain and maintain correction of progressive idiopathic scoliosis. Specifically:

* Diagnosis of idiopathic scoliosis
* Planned recipient of AVBT surgical treatment
* Skeletally immature
* Major Cobb angle ≥30° and ≤65°
* Osseous structure dimensionally adequate to accommodate screw fixation, as determined by radiographic imaging
* Failed or intolerant to bracing

Exclusion Criteria:

* Presence of any systemic infection, local infection, or skin compromise at the anticipated surgical site
* Prior spinal surgery at the level(s) to be treated
* Evidence of documented poor bone quality
* Any other medical or surgical condition which would preclude the potential benefit of spinal surgery, such as coagulation disorders, allergies to the implant materials, and patient's unwillingness or inability to cooperate with post-operative care instructions as determined by the treating physician
* Unwillingness, inability, or living situation (e.g. custody arrangements, homelessness, detention) that would preclude ability to return to the study site for follow-up visits as described in protocol and Informed Consent
* Unwillingness to sign Informed Consent Form and participate in study procedures

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 106 (Estimated)
Dates: Start 2021-09-09 (Actual); Primary Completion 2028-09 (Estimated); Study Completion 2029-09 (Estimated)

PRIMARY OUTCOMES:
The effect on three-dimensional spine growth as compared to normal controls | 5 years
  The three-dimensional spine growth of the subjects will be measured at each study timepoint and compared to known normal controls.
Maintenance of major Cobb angle less than or equal to 50 degrees at skeletal maturity | 5 years
  Subjects who maintain a major Cobb angle less than or equal to 50 degrees at skeletal maturity will be considered a "success."
Complications associated with both the procedure and the device | 5 years
  Subjects will be monitored for complications associated with both the procedure and the device.

CONTACTS AND LOCATIONS:
Overall Officials: Ron El-Hawary, MD, Principal Investigator — Dalhousie University
Locations (12):
- United States (11):
  - Children's National Hospital, Washington D.C., District of Columbia
  - Shriners Children's Chicago, Chicago, Illinois
  - Gillette Children's Specialty Healthcare, Saint Paul, Minnesota
  - Washington University, St Louis, Missouri
  - Morgan Stanley Childrens Hospital of New York-Presbyterian, New York, New York
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Shriners Children's Portland, Portland, Oregon
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - The Medical University of South Carolina, Charleston, South Carolina
  - Vanderbilt University, Nashville, Tennessee
  - Primary Children's Hospital, Salt Lake City, Utah
- Children's Hospital of Eastern Ontario, Ottawa, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Coghlan RF, Oberdorf JA, Sienko S, Aiona MD, Boston BA, Connelly KJ, Bahney C, LaRouche J, Almubarak SM, Coleman DT, Girkontaite I, von der Mark K, Lunstrum GP, Horton WA. A degradation fragment of type X collagen is a real-time marker for bone growth velocity. Sci Transl Med. 2017 Dec 6;9(419):eaan4669. doi: 10.1126/scitranslmed.aan4669. PMID 29212713
- [Background] Trobisch P, Suess O, Schwab F. Idiopathic scoliosis. Dtsch Arztebl Int. 2010 Dec;107(49):875-83; quiz 884. doi: 10.3238/arztebl.2010.0875. Epub 2010 Dec 10. PMID 21191550
- [Background] Karol LA, Johnston C, Mladenov K, Schochet P, Walters P, Browne RH. Pulmonary function following early thoracic fusion in non-neuromuscular scoliosis. J Bone Joint Surg Am. 2008 Jun;90(6):1272-81. doi: 10.2106/JBJS.G.00184. PMID 18519321
- [Background] Samdani AF, Ames RJ, Kimball JS, Pahys JM, Grewal H, Pelletier GJ, Betz RR. Anterior vertebral body tethering for immature adolescent idiopathic scoliosis: one-year results on the first 32 patients. Eur Spine J. 2015 Jul;24(7):1533-9. doi: 10.1007/s00586-014-3706-z. Epub 2014 Dec 16. PMID 25510515
- [Background] Crawford CH 3rd, Lenke LG. Growth modulation by means of anterior tethering resulting in progressive correction of juvenile idiopathic scoliosis: a case report. J Bone Joint Surg Am. 2010 Jan;92(1):202-9. doi: 10.2106/JBJS.H.01728. No abstract available. PMID 20048114
- [Background] Samdani AF, Ames RJ, Kimball JS, Pahys JM, Grewal H, Pelletier GJ, Betz RR. Anterior vertebral body tethering for idiopathic scoliosis: two-year results. Spine (Phila Pa 1976). 2014 Sep 15;39(20):1688-93. doi: 10.1097/BRS.0000000000000472. PMID 24921854
- [Background] Miyanji F, Pawelek J, Nasto LA, Rushton P, Simmonds A, Parent S. Safety and efficacy of anterior vertebral body tethering in the treatment of idiopathic scoliosis. Bone Joint J. 2020 Dec;102-B(12):1703-1708. doi: 10.1302/0301-620X.102B12.BJJ-2020-0426.R1. PMID 33249889
- [Background] Spurway AJ, Hurry JK, Gauthier L, Orlik B, Chukwunyerenwa CK, Kishta WE, El-Hawary R. Three-dimensional True Spine Length: A Novel Technique for Assessing the Outcomes of Scoliosis Surgery. J Pediatr Orthop. 2017 Dec;37(8):e631-e637. doi: 10.1097/BPO.0000000000001031. PMID 28614286
- [Background] Sarwahi V, Wendolowski S, Gecelter R, Maguire K, Gambassi M, Orlando D, Lo Y, Amaral T. When Do Patients Return to Physical Activities and Athletics After Scoliosis Surgery?: A Validated Patient Questionnaire Based Study. Spine (Phila Pa 1976). 2018 Feb 1;43(3):167-171. doi: 10.1097/BRS.0000000000002284. PMID 28604495